CLINICAL TRIAL: NCT02553720
Title: Aquatic Therapy to Lower Adverse and Negative Effects of Venous Thrombosis and InSufficiency
Brief Title: The ATLANTIS Trial
Acronym: ATLANTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona Cardiovascular Consultants (Other)
Collaborators: A.T. Still University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mohsen Sharifi MD, principal investigator, Arizona Cardiovascular Consultants
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ArizonaCC
Record Dates: First submitted 2015-09-10; First posted 2015-09-18 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Chronic Venous Hypertension Due to Deep Vein Thrombosis; Venous Reflux
Keywords: Post thrombotic syndrome; Chronic venous insufficiency
MeSH Terms: conditions — Postthrombotic Syndrome | interventions — Exercise; Water

STUDY DESIGN:
Intervention Model Description: A total of 201 patients were randomized with 100 to the Aquatic Group and 101 to the Control Group. At 24 months, 91 patients had completion of evaluation in the Aquatic Group and 90 patients in the Control Group.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aquatic Group (Experimental): Conventional management plus aquatic exercise At least 15 minutes of walking 3 times/week for 3 months
  Interventions: Other: exercise in water; Other: aquatic activity plus conventional management
- Control Group (Other): Conventional management without aquatic exercise
  Interventions: Other: aquatic activity plus conventional management

INTERVENTIONS:
Other: exercise in water — The patients will be instructed to perform walking or swimming for 15 minutes, 3 times a week for 3 months in a swimming pool in addition to conventional management
  Other Names: aquatic activity
  Arms: Aquatic Group
Other: aquatic activity plus conventional management — walking in water or swimming for 15 minutes, 3 times a week for 3 months in a swimming pool in addition to conventional management

SUMMARY:
The purpose of this study is to test whether addition of aquatic exercise to conventional treatment helps reduce the adverse outcomes of chronic venous insufficiency including CVI resulting from venous thrombosis.

DETAILED DESCRIPTION:
Post-thrombotic syndrome (PTS) develops in approximately 25-60% of patients with acute lower extremity deep venous thrombosis (DVT) depending on severity, chronicity, anatomic level of involvement and efficacy of anticoagulation.The frequency increases with occlusive iliac venous thrombosis. PTS results in significant morbidity and a staggering toll on health careresources . PTS is reduced by early percutaneous endovenous intervention and administration of new oral anticoagulants. There are conflicting results on the efficacy of exercise . In general, exercise has been useful in activation of the muscle pump and improvement of symptoms. There are no data about exercise in a swimming pool. Both walking in water or swimming reduce the effect of joint contact and therefore pain which is particularly useful in patients with arthritis or heavyweight. Furthermore with less effect of gravity, absorption of dependent edema would be faster. Dry skin becomes hydrated and the chlorine of water can exert antiseptic properties. There are no data on the role of aquatic activity in the reduction of measures of venous insufficiency.The purpose of this study is to assess whether encouragement of patients to perform aquatic activity in addition to baseline treatment would positively impact chronic venous insufficiency.

ELIGIBILITY:
Inclusion Criteria:

age>18 years; a Villalta score of ˃5 or a modified Venous Clinical Severity Score (VCSS) of ˃5 plus ongoing symptoms of ˃3 months despite receiving conservative management (minimum of 2 of the following: compression stockings, leg elevation, physical activity on land and use of non-steroidal anti-inflammatory drugs where appropriate, for the preceding 3 months).

Exclusion criteria consisted of unwillingness or inability to use or no access to a swimming pool; open ulceration; planned intervention for arterial or superficial venous reflux, deep venous thrombosis (DVT), venous stenosis, pelvic congestion syndrome, within the first 3 months of enrolment; or using a swimming pool on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
4 point drop in modified VCSS | 3 months and 2 years
  Modified VCSS score at baseline, 3 m and 2 years.

SECONDARY OUTCOMES:
Viallta Score | 3 months and 2 years
  Changes in the Vllalta scoring system
Mortality | 2 years
  Development of death at follow up.
VEINES QOL/Sym | 3months and 2 years
  changes of time velocity integral of the spectral Doppler waveform.
Recurrent venous thromboembolic disease | 3 months and 2 years
  Measured objectively by venous duplex or CT angiography or V/Q scan if indicated
Modified Venous Clinical Severity Score | 3months and 2 years
  Changes in absolute scores before and after intervention
SF 36 questionnaire-PHC | 3 months and 2 years
  Changes in score before and after intervention
Thigh and leg circumference | 3 months and 2 years
  Changes in circumference before and after intervention
"Subjective Index" alteration | 3 months and 2 years
  Changes in score before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen SHARIFI, M.D., Principal Investigator — Arizona Cardiovascular Consultants
Locations (1):
- Arizona cardiovascular consultants, Mesa, Arizona, United States

REFERENCES:
- [Background] Kahn SR, Shapiro S, Ginsberg JS; SOX trial investigators. Compression stockings to prevent post-thrombotic syndrome - Authors' reply. Lancet. 2014 Jul 12;384(9938):130-1. doi: 10.1016/S0140-6736(14)61160-0. No abstract available. PMID 25016993
- [Background] CLOTS (Clots in Legs Or sTockings after Stroke) Trials Collaboration; Dennis M, Sandercock P, Reid J, Graham C, Forbes J, Murray G. Effectiveness of intermittent pneumatic compression in reduction of risk of deep vein thrombosis in patients who have had a stroke (CLOTS 3): a multicentre randomised controlled trial. Lancet. 2013 Aug 10;382(9891):516-24. doi: 10.1016/S0140-6736(13)61050-8. Epub 2013 May 31. PMID 23727163
- [Background] Barwell JR, Davies CE, Deacon J, Harvey K, Minor J, Sassano A, Taylor M, Usher J, Wakely C, Earnshaw JJ, Heather BP, Mitchell DC, Whyman MR, Poskitt KR. Comparison of surgery and compression with compression alone in chronic venous ulceration (ESCHAR study): randomised controlled trial. Lancet. 2004 Jun 5;363(9424):1854-9. doi: 10.1016/S0140-6736(04)16353-8. PMID 15183623
- [Result] Sharifi M, Bay C, Mehdipour M, Sharifi J; TORPEDO Investigators. Thrombus Obliteration by Rapid Percutaneous Endovenous Intervention in Deep Venous Occlusion (TORPEDO) trial: midterm results. J Endovasc Ther. 2012 Apr;19(2):273-80. doi: 10.1583/11-3674MR.1. PMID 22545895